CLINICAL TRIAL: NCT02896309
Title: The Effect of Correction of Metabolic Acidosis in CKD on Intrarenal RAS Activity
Acronym: BIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Ewout Hoorn, Internist nephrologist, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL44415.078.13
Record Dates: First submitted 2016-08-18; First posted 2016-09-12 (Estimated); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Sodium Bicarbonate; Sodium Chloride

ARMS (3):
- Sodium bicarbonate (Experimental): Oral sodium bicarbonate tablets three times daily 1000mg
  Interventions: Dietary Supplement: Sodium bicarbonate
- Sodium chloride (Active Comparator): Oral sodium chloride capsules two times daily 1000mg
  Interventions: Dietary Supplement: Sodium chloride
- No treatment (No Intervention): No treatment

INTERVENTIONS:
Dietary Supplement: Sodium bicarbonate
  Arms: Sodium bicarbonate
Dietary Supplement: Sodium chloride
  Arms: Sodium chloride

SUMMARY:
This study evaluates the effect of oral sodium bicarbonate treatment on the intrarenal renin-angiotensin-system in adult patients with a metabolic acidosis and chronic kidney disease. This treatment is compared to sodium chloride treatment, which serves as control for increased sodium-intake and no treatment, which serves as time-control.

DETAILED DESCRIPTION:
In chronic kidney disease (CKD), as glomerular filtration rate decreases, excretion of hydrogen ions fails, leading to progressive metabolic acidosis (arterial pH < 7.35 and a serum bicarbonate concentration < 22 meq/L). Metabolic acidosis enhances further progression of CKD. It is known that the intrarenal renin-angiotensin system (RAS) is stimulated during metabolic acidosis, but it's specific role in the renal response on changes in the acid-base balance is unknown. Correction of metabolic acidosis by administration of bicarbonate is a common intervention in patients with metabolic acidosis due to chronic kidney disease. It is proven to slow down progression of CKD. There is no knowledge on the effect this therapy has on the intrarenal RAS. Since acidosis does not change serum renin levels, and bicarbonate therapy has no effect on blood pressure, it seems to have no effect on the systemic RAS. The investigators hypothesize that bicarbonate therapy diminishes intrarenal RAS activity without affecting the systemic RAS.

ELIGIBILITY:
Inclusion Criteria:

* male or female adult (≥18 years)
* chronic kidney disease stage 4, i.e. estimated glomerular filtration rate (MDRD) 15-30 ml/min
* plasma bicarbonate concentration of 15-24 meq/L

Exclusion Criteria:

* bicarbonate level >24 meq/L or <15 meq/L, the latter because in that case it seems highly recommended to start sodium bicarbonate suppletion and not to postpone this
* sodium bicarbonate use in the 1 month preceding the study
* heart failure
* liver cirrhosis
* blood pressure >140/90 mmHg despite the use of 3 different antihypertensives
* a kidney transplant in situ
* a history of nonadherence to medication
* use of calcineurin inhibitors (these immunosuppressive drugs are known to induce metabolic acidosis and influence electrolytes and acid-base balance)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2018-12-27 (Actual)

PRIMARY OUTCOMES:
Urinary renin concentration | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ewout J Hoorn, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Background] de Brito-Ashurst I, Varagunam M, Raftery MJ, Yaqoob MM. Bicarbonate supplementation slows progression of CKD and improves nutritional status. J Am Soc Nephrol. 2009 Sep;20(9):2075-84. doi: 10.1681/ASN.2008111205. Epub 2009 Jul 16. PMID 19608703
- [Background] Ng HY, Chen HC, Tsai YC, Yang YK, Lee CT. Activation of intrarenal renin-angiotensin system during metabolic acidosis. Am J Nephrol. 2011;34(1):55-63. doi: 10.1159/000328742. Epub 2011 Jun 10. PMID 21659740
- [Background] Nagami GT. Role of angiotensin II in the enhancement of ammonia production and secretion by the proximal tubule in metabolic acidosis. Am J Physiol Renal Physiol. 2008 Apr;294(4):F874-80. doi: 10.1152/ajprenal.00286.2007. Epub 2008 Feb 20. PMID 18287403
- [Background] Henger A, Tutt P, Riesen WF, Hulter HN, Krapf R. Acid-base and endocrine effects of aldosterone and angiotensin II inhibition in metabolic acidosis in human patients. J Lab Clin Med. 2000 Nov;136(5):379-89. doi: 10.1067/mlc.2000.110371. PMID 11079465